CLINICAL TRIAL: NCT07268807
Title: Effect of Roxadustat on Heart Failure Patients With Anaemia and Moderate-to-Severe Chronic Kidney Disease: A Single-Centre Retrospective Study
Brief Title: Effect of Roxadustat on Heart Failure Patients With Anaemia and Moderate-to-Severe Chronic Kidney Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Zhongda Hospital (Other)
Responsible Party: Principal Investigator, Wenbin Lu, associate chief physician; Associate Professor, Zhongda Hospital
Other Study IDs: 2025ZDSYLL380-P01
Record Dates: First submitted 2025-11-14; First posted 2025-12-08 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-09

CONDITIONS: Heart Failure; CKD; Anemia
MeSH Terms: conditions — Heart Failure; Anemia | interventions — roxadustat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- treated with Roxadustat
  Interventions: Drug: Roxadustat
- No treated with HIF-PHIs

INTERVENTIONS:
Drug: Roxadustat — treated by Roxadustat
  Groups: treated with Roxadustat

SUMMARY:
Previous clinical observations of potential benefit from Roxadustat in this complex patient population prompted this investigation Therefore, the investigators designed this retrospective, observational study to thoroughly investigate the effects of Roxadustat on heart failure treatment and ventricular remodelling in this specific patient population, aiming to provide new insights for patients management.

ELIGIBILITY:
Inclusion Criteria:

* aged 18-85 years, regardless of gender;
* fulfilled the diagnostic criteria for heart failure and chronic kidney disease;
* haemoglobin level <130 g/L for men or <120 g/L for women at baseline;
* had regularly received Roxadustat for over one year;
* possessed complete clinical data, including information from pre-specified time points.

Exclusion Criteria:

* comorbid myelodysplastic syndromes, multiple myeloma, hereditary hematologic diseases (e.g., thalassemia, sickle cell anaemia, pure red cell aplasia), hemosiderosis, hemochromatosis, or other disorders confirmed to cause anaemia due to erythrocyte destruction and/or abnormal hematopoietic function;
* haemoglobin level ≤45 g/L on two or more blood tests, a history of major bleeding within one year, or a history of anaemia corrected by blood transfusion;
* bilateral nephrectomy, kidney transplantation within ≤6 months, or congenital kidney diseases (e.g., polycystic kidney disease);
* hypertrophic obstructive cardiomyopathy or congenital heart disease with right-to-left shunt;
* comorbid malignancy with an investigator-assessed life expectancy of less than 12 months;
* pregnancy or lactation;
* known allergy to the study drug (active ingredient or excipients);
* participation in a drug clinical trial within one year.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Heart Failure Patients with Anaemia and Moderate-to-Severe Chronic Kidney Disease
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2026-09-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Mace | 1 year
  MACE was defined as the occurrence of any of the following: all-cause mortality, hospitalization for unstable angina or coronary revascularization, heart failure rehospitalization, or ischemic stroke.
BNP | 1 year
  B-type natriuretic peptide
NYHA functional classification | 1 year
  I: No limitation of physical activity. Ordinary physical activity does not cause undue fatigue, palpitation or shortness of breath.
  II: Slight limitation of physical activity. Comfortable at rest. Ordinary physical activity results in fatigue, palpitation, shortness of breath or chest pain.
  III: Marked limitation of physical activity. Comfortable at rest. Less than ordinary activity causes fatigue, palpitation, shortness of breath or chest pain.
  IV: Symptoms of heart failure at rest. Any physical activity causes further discomfort.
left ventricular ejection fraction (LVEF) | 1 year
left ventricular end-diastolic dimension (LVEDD) | 1 year
interventricular septal thickness (IVS) | 1 year
left ventricular posterior wall thickness (LVPW) | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongda hospital Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided
No application for disclosure has been submitted to the Clinical Ethics Committee.

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan: Version 1.0.1 (2025-12-03): https://cdn.clinicaltrials.gov/large-docs/07/NCT07268807/Prot_SAP_000.pdf
  • Study Protocol and Statistical Analysis Plan: Version 1.0.0 (2025-09-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT07268807/Prot_SAP_001.pdf
  • Study Protocol and Statistical Analysis Plan: No cover page (2025-09-01): https://cdn.clinicaltrials.gov/large-docs/07/NCT07268807/Prot_SAP_002.pdf